CLINICAL TRIAL: NCT02863016
Title: tHe Effects of Postdilution Online Hemodiafiltration With AcEtate-free Citrate dialySis Fluid on Inflammation Markers in TUscan Prevalent Hemodialysis patientS: HEPHAESTUS Study
Brief Title: Effects of Postdilution Online Hemodiafiltration With AcEtate-free Citrate dialySis Fluid on Inflammation Markers
Acronym: HEPHAESTUS
Status: Completed | Type: Observational
Sponsor: Ospedale Santa Maria Annunziata (Other)
Responsible Party: Principal Investigator, Francesco Pizzarelli, Principal Investigator, Ospedale Santa Maria Annunziata
Other Study IDs: HEPHAESTUS_020713
Record Dates: First submitted 2016-08-01; First posted 2016-08-11 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: ESRD
Keywords: dialysis; hemodiafiltration
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Concentrate SelectBag One: Each patient will be subjected to two stages of each month, where it will be treated with online HDF postdilution: first of all concentrate SelectBag One (with 3 mM of acetic acid and 0 mM of citrate)
  Interventions: Device: SelectBag One
- Concentrate SelectBag Citrate: Each patient will be subjected to two stages of each month, where it will be treated with online HDF postdilution, then with SelectBag Citrate (with 0 mM of acetic acid and 1 mM of citric acid)
  Interventions: Device: SelectBag One

INTERVENTIONS:
Device: SelectBag One — Each patient will be subjected to two stages of each month, where it will be treated with online HDF postdilution with two kind of concentrates: acetic acid (Ac-HDF) and acetate-free citrate containing one (HDF-Cit ). For each of the sessions will be used online HDF postdilution with TMP biofeedback (UltraControl) and Filter high permeability.
  Other Names: SelectBag Citrate

SUMMARY:
The aim of this study was to evaluate the effect and timing of action on the inflammatory state of a acetate-free containing citrate concentrate (Cit-, 1 mM Citrate) in online postidultion HDF with high volumes compared to traditional concentrated (Ac-, 3 mM of acetate ) in the medium term. In addition, the study will evaluate other parameters of efficiency dialysis, cardiovascular stability, the safety of the concentrate with regard to bone metabolism and vessel calcification in the medium term.

DETAILED DESCRIPTION:
The primary objective of this study was to evaluate if a hemodiafiltration with concentrated citrate (Cit-HDF) in 3 months can reduce the inflammation markers, evaluated by a Predialytic value of Beta2-microglobulin (B2m), CRP and IL6 compared to traditional concentrated acetic acid (Ac-HDF).

The secondary objectives of this study are to evaluate if Cit-HDF, compared to Ac-HDF, can have an effect in a period of 3 months on the following aspects:

* the change weekly pre-dialysis values of other markers of oxidative stress (TAC, NF-kB);
* the technical parameters of HDF treatment, such as convective volumes, and blood pressure in the circuit in the filter (TMP, pressure pre-filter);
* the cardiovascular stability through blood pressure and heart rate before and after dialysis (SBP, DBP, HR) and number of intradialytic hypotension;
* the parameters of safety as the variation of the values of the mobility Predialytic bone (PTH, alkaline phosphatase, fetuin-A), the variation of the values intradialytic biochemical impacted by citrate (total and ionized calcium, bicarbonate) and clotting time (aPTT);
* the variation of calcifications observed by:

  * the expression of molecules that express the ability of calcification of muscle cells and endothelial cells in culture with plasma taken at the beginning of treatment
  * a measure of carotid intimal thickness and pulse vawe velocity by Eco Color Doppler (optional);
* dialysis efficiency by varying pre-and post-dialysis (RR%) and Clearance average molecular weight solutes with small and medium (Phosphorus, Beta2 Micro, Myoglobin) and indices of dialysis adequacy of small molecules such as EKT / V based on the dialysance ion formula Watson (calculated automatically by the monitor to dialysis);

ELIGIBILITY:
Inclusion Criteria:

. Patients clinically stable.

* age> 18.
* HDF in renal replacement therapy for more than 1 month.
* good functionality of the vascular blood flow that allows real at least 250 ml / min. and recirculation below 10%.

Exclusion Criteria:

* Life expectancy <3 months.
* With residual renal function> 500 ml / day.
* Vascular access with CVC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Patients clinically stable.
  * age> 18.
  * HDF in renal replacement therapy for more than 1 month.
  * good functionality of the vascular blood flow that allows real at least 250 ml / min. and recirculation below 10%.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Inflammation | 3 months
  Value of IL-6

SECONDARY OUTCOMES:
Dialytic dose | 3 months
  convective exchange volumes

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Pizzarelli, Dr, Principal Investigator — Ospedale Santa Maria Annunziata_ Firenze (Italy)
Locations (3):
- Italy (3):
  - Ospedale Santa Maria Annunziata, Florence, Fi
  - Ospedale Versilia, Lido di Camaiore, Lucca
  - Ospedale Campo di Marte, Lucca

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maduell F, Moreso F, Pons M, Ramos R, Mora-Macia J, Carreras J, Soler J, Torres F, Campistol JM, Martinez-Castelao A; ESHOL Study Group. High-efficiency postdilution online hemodiafiltration reduces all-cause mortality in hemodialysis patients. J Am Soc Nephrol. 2013 Feb;24(3):487-97. doi: 10.1681/ASN.2012080875. Epub 2013 Feb 14. PMID 23411788
- [Background] Panichi V., Bernabini G., Fanelli R., Rosati A., Pizzarelli F. Emodiafiltrazione (HDF) on line in post-diluizione con un nuovo concentrato acido a base di citrato: risultati di uno studio pilota multicentrico. Atti Convegno SIN, Genova, 2011
- [Background] Matsuyama K, Tomo T, Kadota J. Acetate-free blood purification can impact improved nutritional status in hemodialysis patients. J Artif Organs. 2011 Jun;14(2):112-9. doi: 10.1007/s10047-010-0551-7. Epub 2011 Feb 19. PMID 21336818
- [Derived] Pizzarelli F, Cantaluppi V, Panichi V, Toccafondi A, Ferro G, Farruggio S, Grossini E, Dattolo PC, Miniello V, Migliori M, Grimaldi C, Casani A, Borzumati M, Cusinato S, Capitanini A, Quercia A, Filiberti O, Dani L; Hephaestus study group. Citrate high volume on-line hemodiafiltration modulates serum Interleukin-6 and Klotho levels: the multicenter randomized controlled study "Hephaestus". J Nephrol. 2021 Oct;34(5):1701-1710. doi: 10.1007/s40620-020-00943-6. Epub 2021 Feb 9. PMID 33559851